CLINICAL TRIAL: NCT04342247
Title: Effects of External Testosteron Intake on the Choroid: Enhance-depth Imaging Optical
Brief Title: Effects of External Testosteron Intake on the Choroid: Enhance-depth Imaging Optical Coherence Tomography Study
Status: Completed | Type: Observational
Sponsor: Neon Hospital (Other)
Responsible Party: Principal Investigator, Volkan YETER, Asistan of Professor, Ondokuz Mayıs University
Other Study IDs: 2019/568
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Effects of the External Testosteron Intake Over the Choroids of the Patients With Androgen Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- androgen deficient
  Interventions: Drug: external testosteron
- healthy

INTERVENTIONS:
Drug: external testosteron — external testosteron
  Groups: androgen deficient

SUMMARY:
According to the results Ciloğlu et al., CSC is related to elevated total testosterone levels. Testosterone may play a role in predisposing males to CSC. Thus, we aimed to investigate the possible effect of external testosteron intake over choroidal parameters; such as choroidal thickness, choroidal vascularity index, choroidal stromal ve luminal areas,ect.

DETAILED DESCRIPTION:
In the study, we have two group: First group consists of patients with testosteron deficiency and there are sex and age-matched healthy control subjects in the second group. We will measure the parameters of both groups at baseline. And first month and 3rd month we will remeasure the values of the parameters by enhance depth optical coherence tomography. The results will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

for androgen deficient group: no other ocular and systemic disease except androgen deficiency. no history of ocular surgery or disease no medicine use for healthy controls :no other ocular and systemic disease. no history of ocular surgery or disease no medicine use, no smoking or any tobocco use

Exclusion Criteria:having any ocular and systemic disease. history of ocular surgery or disease,medicine use, smoking or any tobocco use

-

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: randomly selected subjects aged between 30 and 800
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
to evaluate Effects of External Testosteron Intake on the Choroid: Enhance-depth Imaging Optical Coherence Tomography Study | 2019 and 20120
  to obtain the measurements of the choroids

CONTACTS AND LOCATIONS:
Locations (1):
- Volkan YETER, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No